CLINICAL TRIAL: NCT06734546
Title: The Effect of Exercise of High Vs. Moderate Intensity on the Brain in Type 2 Diabetes
Brief Title: The Effect of Exercise on the Brain in Type 2 Diabetes
Acronym: SAINT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Jessa Hospital (Other); Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Full professor, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B1152024000012; 1129225N (Other Grant/Funding Number: FWO (Fonds Wetenschappelijk Onderzoek)); BOF24KP05 (Other Grant/Funding Number: BOF (Bijzonder Onderzoeksfonds))
Record Dates: First submitted 2024-11-25; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; exercise intervention; brain; cognition; neurometabolism; dementia; cerebral perfusion
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High intensity exercise training group (Experimental): This arm will receive 6 months of exercise training at high intensity (105% VT2)
  Interventions: Other: Exercise intervention
- Moderate intensity exercise training group (Experimental): This arm will receive 6 months of exercise training at moderate intensity (60% VT2)
  Interventions: Other: Exercise intervention
- Control group (No Intervention): This arm won't receive exercise training

INTERVENTIONS:
Other: Exercise intervention — The exercise intervention entails 6 months of supervised exercise on a hometrainer at high or moderate intensity, 3 times per week
  Arms: High intensity exercise training group; Moderate intensity exercise training group

SUMMARY:
The goal of this clinical trial is to learn if exercise training of high or moderate intensity is most optimal to improve brain health and prevent neurodegeneration in type 2 diabetes patients. The main question it aims to answer is:

What is the effect of exercise training of high vs. moderate intensity on brain metabolism, brain perfusion, and cognition in type 2 diabetes?

Researchers will compare the exercise training groups to a control group without exercise training to determine the effect of exercise training on the brain in type 2 diabetes.

Participants will exercise for 6 months, 3 times per week. Before and after these 6 months, they will undergo:

* a brain MRI scan
* cognitive tests
* blood sampling

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* no insulin therapy
* 30-75 years old
* right handed
* physically inactive

Exclusion Criteria:

* left handed
* MRI contraindications
* psychological disorders
* exogenous insulin therapy
* history of coma, transient ischemic attack, head trauma, brain tumor, stroke, epilepsy, and other central nervous system diseases that could cause dementia or presence of dementia before T2DM
* suffering from any disease with significant impact on exercise intervention participation such as: chronic heart disease (e.g. valve insufficiency ≥ grade 2) or significant arrhythmias, cardiac events less than one year ago (myocardial infarction, coronary artery bypass graft, percutaneous coronary intervention), clinical heart failure (oedema, shortness of breath), percutaneous coronary intervention less than one year ago, chronic obstructive pulmonary disease (COPD), cerebrovascular or peripheral vascular disease
* severe hypertension (>160/110 mmHg)
* ongoing cancer, severe neuropathy (limiting exercise participation)
* renal disease (GRF <45 ml/min/1,73 m2)
* inability to regularly participate in the exercise intervention
* pregnancy
* breastfeeding

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Neurometabolite levels | From enrollment to the end of treatment at 6 months
  Levels of N-acetylaspartate, choline, myo-inositol, creatine, glutathion, and glutamate, measured in institutional units (i.u.) by means of magnetic resonance spectroscopy (MRS).
Changes in arterial spin labelling measured by means of magnetic resonance imaging (MRI) | From enrollment to the end of treatment at 6 months
  Changes in cerebral perfusion expressed in mL/100g/min, and blood flow through the blood-brain-barrier expressed in milliseconds

SECONDARY OUTCOMES:
Levels of neurodegenerative blood biomarkers | From enrollment to the end of treatment at 6 months
  Tau (pg/mL), amyloid beta (pg/mL), S100B (ng/mL), neurofilament light (pg/mL) etc.
Blood lipid profile | From enrollment to the end of treatment at 6 months
  This outcome measure includes assessments of the lipid profile, reported in milligrams per deciliter (mg/dL) or millimoles per liter (mmol/L):
  High-Density Lipoprotein (HDL), Low-Density Lipoprotein (LDL), Triglycerides, Free Fatty Acids, Total Cholesterol
Brain volume | From enrollment to the end of treatment at 6 months
  Total and regional (LHIPP, mPFC, PCC) brain volumes
Diffusion-weighted magnetic resonance imaging | From enrollment to the end of treatment at 6 months
  DWI will be used to measure differences in Brownian motion of water molecules within the brain
Fasted blood glucose | From enrollment to the end of treatment at 6 months
  Fasting Glucose: Reported in milligrams per deciliter (mg/dL) or millimoles per liter (mmol/L).
Kidney function (eGFR) | From enrollment to the end of treatment at 6 months
  Estimated Glomerular Filtration Rate (eGFR): Reported in milliliters per minute per 1.73 m² (mL/min/1.73 m²).
Cognitive function: MoCA | From enrollment to the end of treatment at 6 months
  Cognitive function as assessed by the Montreal Cognitive Assessment (MoCA), scored on a scale of 0-30.
Cognitive function: Face recognition test | From enrollment to the end of treatment at 6 months
  Cognitive function as assessed by the Face Recognition Test, reported as the number of correct identifications.
Cognitive function: Object location test | From enrollment to the end of treatment at 6 months
  Cognitive function as assessed by the Object Location Test, reported as the number of correct placements.
Cognitive function: Trail making test | From enrollment to the end of treatment at 6 months
  Cognitive function as assessed by the Trail Making Test, reported as time to completion (seconds) for Parts A and B.
Cognitive function: Stroop colour and word test | From enrollment to the end of treatment at 6 months
  Cognitive function as assessed by the Stroop Color and Word Test, reported as time to completion (seconds) or number of errors.
Cognitive function: Rey auditory verbal learning test | From enrollment to the end of treatment at 6 months
  Cognitive function as assessed by the Rey Auditory Verbal Learning Test, reported as the number of words recalled.
Subjective cognitive function | From enrollment to the end of treatment at 6 months
  Cognitive function as assessed by the Cognitive Failure Questionnaire, scored on a scale of 0-100.
Peak load during CPET | From enrollment to the end of treatment at 6 months
  The maximum load achieved during cardiopulmonary exercise testing (CPET) on a bicycle, measured in watts.
VO2peak during CPET | From enrollment to the end of treatment at 6 months
  The peak oxygen consumption measured during CPET, indicating the maximal capacity for oxygen utilization during exercise.
  Unit of Measure: Milliliters per kilogram per minute (mL/kg/min).
Fasted blood HbA1c | From enrollment to the end of treatment at 6 months
  Hemoglobin A1c (HbA1c): Reported as a percentage (%).
Fasting insulin | From enrollment to the end of treatment at 6 months
  Fasting Insulin: Reported in micro-international units per milliliter (μIU/mL) or picomoles per liter (pmol/L).
Kidney function (creatinine) | From enrollment to the end of treatment at 6 months
  Creatinine: Reported in milligrams per deciliter (mg/dL) or micromoles per liter (μmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hansen, Full professor, Principal Investigator — Hasselt University; Koen Cuypers, Assistant professor, Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided